CLINICAL TRIAL: NCT00021320
Title: Phase II Evaluation Of Paclitaxel, Cisplatin And 5-Fluorouracil Given In Combination With Radiation Therapy Prior To Surgery In Patients With Resectable Esophageal Cancer
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068769; P30CA006927 (NIH); FCCC-00003; NCI-G01-1982
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Esophageal Cancer
Keywords: stage 0 esophageal cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Fluorouracil; Paclitaxel; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: paclitaxel
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with or without radiation therapy in treating patients who have esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the median and two-year disease-free and overall survival of patients with resectable esophageal cancer treated with neoadjuvant paclitaxel, cisplatin, and fluorouracil with concurrent radiotherapy.
* Determine the complete and partial responses in patients treated with this regimen.
* Assess the toxicity of this regimen in these patients.
* Determine the optimal dose of paclitaxel when administered in this regimen in these patients.
* Determine the effect of tumor tubulin isoform expression on chemosensitivity and overall survival of patients treated with this regimen.

OUTLINE: Patients receive paclitaxel IV over 3 hours and cisplatin IV over 1 hour on day 1. Treatment repeats every 3 weeks for 2 courses.

Beginning 3 weeks after completion of initial chemotherapy, patients receive concurrent chemoradiotherapy comprising paclitaxel IV over 1 hour and cisplatin IV over 1 hour on days 1, 8, 15, 22, and 29; fluorouracil IV continuously for 5 weeks; and radiotherapy daily 5 days a week for 5 weeks.

At 4-8 weeks after completion of chemoradiotherapy, patients may undergo surgical resection. Patients with local progressive disease after 2 courses of initial chemotherapy undergo surgical resection instead of receiving concurrent chemoradiotherapy.

Patients are followed within 6 weeks, every 3 months for 3 years, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma, squamous cell, adenosquamous, or undifferentiated carcinoma of the esophagus or gastroesophageal junction

  * Potentially resectable disease
* No malignant celiac node involvement
* No cervical esophageal carcinoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,800/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Other:

* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No significant medical or psychiatric illness that would preclude study
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for at least 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for esophageal cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior thoracic radiotherapy

Surgery:

* See Disease Characteristics
* No prior surgical resection of esophageal tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-05; Primary Completion 2004-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cheng, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States